CLINICAL TRIAL: NCT00953836
Title: Kinetic Study of Two Known Alkylresorcinol Metabolites in Human Subjects After the Intake of Rye Fiber, the Most Abundant Source of Alkylresorcinols in Diet.
Brief Title: Plasma Pharmacokinetics of Alkylresorcinol Metabolites; New Candidate Biomarkers for Whole Grain Rye and Wheat Intake
Acronym: Rye-kinetics
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Samfundet Folkhälsan (Unknown); Sigrid Jusélius Foundation (Other)
Other Study IDs: 22/13/03/00/09
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Kinetics of Alkylresorcinol Metabolites
Keywords: kinetics; alkylresorcinol metabolites; rye fiber

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to investigate the kinetics of two known alkylresorcinol metabolites in human subjects after intake of high-fiber rye bread. Whole grain rye is the most abundant source of alkylresorcinols.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, volunteer

Exclusion Criteria:

* Hemoglobin below 125 mmol/L in females and below 135 mmol/L in males use of antibiotics within 3 months before entering the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy, free-living females and males
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matti J Tikkanen, M.D., prof., Study Director — Department of Medicine, University of Helsinki, Helsinki, Finland
Locations (1):
- Folkhälsan Research Center, Helsinki, Finland